CLINICAL TRIAL: NCT02048592
Title: Impact of Immunonutrition on the Patients With Cystic Fibrosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Ondrej Hloch MD, Dpt. of of Internal Medicine, 2nd Medical School of Charles Universty and University Hospital Moto, University Hospital, Motol
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: FN Motol-project 6008; EK-942/13 (Other: Faculty hospital Prague Motol)
Record Dates: First submitted 2013-12-16; First posted 2014-01-29 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Cystic Fibrosis; Malnutrition; Oxidative Stress
Keywords: cystic fibrosis, immunonutrition, oxidative stress
MeSH Terms: conditions — Cystic Fibrosis; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Impact-Nutridrink (Active Comparator): The first arm will be given immunonutrition -Impact- for 8 weeks, afterwards the patients will return to their previous nutrition support for another 8 weeks. We expect the improvement of oxidative stress parameters after 8 weeks of immunonutriton and return to baseline values when immunonutrition is stopped
  Interventions: Dietary Supplement: Impact-Nutridrink
- Nutridrink-Impact (Active Comparator): The second group will be given their previous nutrition support (Nutridrink) for 8 weeks, afterwards the patients will be switched to immunonutrition- Impact- for another 8 weeks. In this group of patients we do not expect any change of oxidative stress parameters after the first 8 weeks. The improvement is expected at the end of the second half of study.
  Interventions: Dietary Supplement: Nutridrink-Impact

INTERVENTIONS:
Dietary Supplement: Impact-Nutridrink — IMPACT (immunonutrition) will be given in the first 8 weeks. Afterwards the patients will be returned to their previous nutrition support |(Nutridrink) for another 8 weeks.
  Other Names: Impact is brand name of oral nutrition produced by Nestle-Switzerland. It improves immune system; Nutridrink is brand name of oral nutrition produced by company Nutricia (Denmark) with no effect on immune system.
  Arms: Impact-Nutridrink
Dietary Supplement: Nutridrink-Impact — In this group of patients - the study starts with period of 8 weeks with no change of previous nutrition support (Nutridrink). After 8 weeks the laboratory results will be examined ant the patients will switch to immunonutrition (Impact) for another 8 weeks. After the laboratory examination including oxidative stress parameters will be evaluated.
  Other Names: Impact- brand name for immunonutrition - company Nestle Switzerland; Nutridrink- nutrition of company Nutriticia (Denmark)- with no immune response
  Arms: Nutridrink-Impact

SUMMARY:
The primary objectives:

To evaluate the effect of immunonutrition on the adult patient suffering from cystic fibrosis

1. Safety of immunonutrition
2. The effect of immunonutrition on parameters of oxidative stress
3. The effect of immunonutrition on the inflammatory parameters
4. The effect of immunonutrition on nutrition status

Hypothesis

The high oxidative stress is present in patients with cystic fibrosis. Immunonutrition has been shown to positively modulate oxidative stress in the different clinical setting however it has not yet been evaluated inpatients with cystic fibrosis who frequently need some support by means of enteral nutrition. We anticipate that the substitution of routine enteral nutrition by immunonutrition will result in improving of oxidative stress parameters.

,

DETAILED DESCRIPTION:
Method Crossover open study will take 16 weeks. The patients eligible for the study according to inclusion and exclusion criteria are going to be divided into 2 groups after signing the informed consent. In both groups their nutrition status, humoral and cellular immunity, respiratory system function and parameters of oxidative stress will be evaluated before entering the intervention.

Afterwards the patients are going to be divided into one group who will receive nutrition support using immunonutrition for the next 8 weeks while the second one will continue with their nutrition support using routine sipping support with no immunonutrition. According to our hypothesis oxidative stress parameters will improve in the group of patients on immunonutrition comparing to the other group. Afterwards the patients will change their nutrition support for another 8 weeks. The patients who took immunonutrition in the first half of study will switch back to routine sipping support and contrary the patients who were in the first part of study on routine sipping will take immunonutrition. After the end of this period of study we expect the return of oxidative stress parameters to the baseline values in the group of patients who took immunonutrition in the first half of study but who were returned to routine nutrition support and contrary the improvement of oxidative stress parameters in the patients who started to take immunonutrition in the second half of study.

The total energy support will be identical in both periods for each individual patient. After the first 8 weeks and after the completion of study the same examination are going to be evaluate as it was on the entrance to study.

Statistical analysis: means, SD, t-test, chi square test, Mann Whitney test, linear correlation and multilinear analysis

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis
* adult, elder 18 years
* enteral nutrition at least for the last 12 monthes

Exclusion Criteria:

* patient waiting for lung transplant
* patients with another life limiting disease-e.g. cancers

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
to evaluate the change of oxidative stress in patients with cystic fibrosis induced by immunonutrition | 16 weeks
  Oxidative stress and parameters of antioxidant activity will be evaluated when the nutrition support is provided with classic sipping (Nutridrink-Nutricia) or by immunonutrition (Impact-Nestle)

SECONDARY OUTCOMES:
to evaluate the change of inflammatory parameters in patients with cystic fibrosis induced by the application of immunonutrition | 16 weeks

OTHER OUTCOMES:
to evaluate the change of nutrition parameters in patients with cysic fibrosis induced by the application of immunonutrition | 16 weeks
to evaluate the change of respiratory function in patients with cystic fibrosis induced by immunonutrition | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ondrej Hloch, MD, Principal Investigator — Faculty hospital Motol; Jiri Charvat, MD, Study Chair — Faculty hospital Motol; Milan Kvapil, MD, Study Director — Faculty hospital Motol
Locations (1):
- Faculty hospital Motol, Prague, Czechia